CLINICAL TRIAL: NCT05285436
Title: A Prospective Clinical Study to Assess the Clinical Utility of Turbidity With the CloudCath System in Patients Using In-Home Peritoneal Dialysis
Brief Title: A Prospective Clinical Study to Assess the Clinical Utility of Turbidity in Patients Using In-Home Peritoneal Dialysis
Acronym: ACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CloudCath (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CC-P-002
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: End Stage Renal Disease; Peritoneal Dialysis-associated Peritonitis; Peritonitis
MeSH Terms: conditions — Kidney Failure, Chronic; Peritonitis

STUDY DESIGN:
Intervention Model Description: All study participants receive a CloudCath Device and use it at home adjunctively to their regular peritoneal dialysis system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CloudCath detection (Experimental): Active monitoring of dialysate effluent by the CloudCath System.
  Interventions: Device: CloudCath System

INTERVENTIONS:
Device: CloudCath System — The CloudCath System enables drainage and measures turbidity, reported as a numeric score, in peritoneal dialysate effluent.

SUMMARY:
This study aims to determine if the CloudCath device can detect infections related to peritoneal dialysis (peritonitis) as fast or faster than the current standard methods used by patients and doctors to detect such infections.

DETAILED DESCRIPTION:
This study will evaluate the safety and effectiveness of the CloudCath System to detect the onset of peritonitis as compared to standard of care.

Study Participants will connect the CloudCath System to their home peritoneal dialysis unit and the CloudCath System will analyze the effluent dialysis solution for changes associated with peritonitis. The system will alert the participant and healthcare provider if it detects a possible infection so they can be formally diagnosed by their healthcare provider.

Following enrollment, Study Participants will use the CloudCath System for 12 continuous months.

Study results from the ACT study will be compared to the results of the CATCH Study (Protocol number CC-P-001; NCT04515498). In CATCH, the Study Participants used a CloudCath System; however, the notification capabilities (per the CloudCath System algorithm) were deactivated.

ELIGIBILITY:
Key Inclusion Criteria:

* currently using peritoneal dialysis
* provides informed consent
* willing to comply with the requirements of the study
* has cellular data coverage at home

Key Exclusion Criteria:

* active or history of cancer requiring chemotherapy within prior 6 months
* signs or symptoms of an active infection within 14 days prior to enrollment
* peritonitis diagnosis within 30 days prior to enrollment
* participating in another investigational device or drug study that may potentially affect study results
* other medical, social or psychological problems that, in the opinion of the investigator, exclude the study participant from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time to peritonitis diagnosis | 12-months
  The time between detection by the CloudCath System and laboratory confirmation of peritonitis.

SECONDARY OUTCOMES:
Agreement in peritonitis detection between the CloudCath System and clinical criteria. | 12-months
  clinical criteria include: white blood cells (WBC) (>100 cells per microliter or >0.1 x10^9/L), polymorphonuclear cells (PMN) (>50%), microbiology culture results, gram staining, and peritonitis symptoms
Agreement in detection of clinically actionable events between the CloudCath System and laboratory reports and/or diagnosis | 12-months
  Clinically actionable events defined as an event which requires treatment (i.e., prescribing medications, cleaning an exit site, etc) or intervention (i.e., PD catheter manipulation, removal).
  Events of interest for this protocol include, but are not limited to, peritonitis, exit site or tunnel infection, and peritoneal dialysis (PD) catheter dysfunction (including PD catheter-related bleeding and PD catheter-related drainage issues).
Agreement in detection of clinically relevant events based on CloudCath System, as compared to clinical laboratory results or diagnosis of a clinically relevant event. | 12-months
  Clinically relevant events are defined as clinically actionable events, events treated preventatively or medically relevant events.
Sensitivity and Specificity of the CloudCath System to detect peritonitis as compared to diagnostic laboratory testing | 12-months
  Analysis of sensitivity and specificity of CloudCath System detection of peritonitis, as compared to diagnostic laboratory testing

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Chertow, MD, Study Director — Stanford University
Locations (1):
- Dialysis Center of Western Massachusetts Llc, Chicopee, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No